CLINICAL TRIAL: NCT03895476
Title: A Randomized Controlled Trial to Measure Pain Perception Following De-Epithelized Free Gingival Graft Harvesting
Brief Title: To Measure Pain Perception Following De-Epithelized Free Gingival Graft Harvesting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hussein Basma, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300002777; UAB Periodontology (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Gingival Recession; Palate; Wound
MeSH Terms: conditions — Gingival Recession; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Collagen Plug with sutures (Active Comparator): Palatal wound will be protected with collagen plug and sutures.
  Interventions: Diagnostic Test: palatal wound will be cover with collagen and sutures
- Platelet Rich Fibrin (PRF) (Active Comparator): palatal wound will be protected with Platelet rich Fibrin
  Interventions: Diagnostic Test: palatal wound covered with platelet rich fibrin
- Collagen Plug with Cyanoacrylate (CPC) (Active Comparator): Palatal wound will consist of collagen protection with the additional layer of cyanoacrylate surgical glue.
  Interventions: Diagnostic Test: palatal wound covered with a collagen sponge and cyanoacrylate
- Palatal Stent (Active Comparator): Palatal wound will be protected with palatal stent.
  Interventions: Diagnostic Test: palatal wound covered with a stent

INTERVENTIONS:
Diagnostic Test: palatal wound will be cover with collagen and sutures — after harvesting the graft from the palate, a collagen sponge will be sutured to cover the harvested site
  Arms: Collagen Plug with sutures
Diagnostic Test: palatal wound covered with platelet rich fibrin — after harvesting the graft from the palate the platelet rich fibrin will be sutured to covered the harvested site
  Arms: Platelet Rich Fibrin (PRF)
Diagnostic Test: palatal wound covered with a collagen sponge and cyanoacrylate — after harvesting the graft from the palate a collagen sponge will be sealed with cyanoacrylate in position
  Arms: Collagen Plug with Cyanoacrylate (CPC)
Diagnostic Test: palatal wound covered with a stent — after harvesting the graft from the palate a stent that will be prepared for the patient, will be placed on to cover the wound
  Arms: Palatal Stent

SUMMARY:
This randomized clinical comparative study will evaluate the postoperative pain following the FGG graft harvest procedure technique covered by four different methods for coverage of the palatal donor site.

DETAILED DESCRIPTION:
This study will compare the application of :

* hemostatic collagen sponge
* collagen sponge sealed with abio-adhesive material
* Platelet rich fibrin
* physical barrier (stent) on the palatal donor sites with the purpose of which one of these will result in least postoperative pain after epithelialized gingival graft (EGG) harvesting.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old- 70 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* Patients needing soft tissue graft with teeth that have miller class I or II recession (>=2mm) on the facial aspects
* Presence of periodontally healthy teeth at the recipient site.
* Ability of the participants to maintain good oral hygiene
* Patient not pregnant or breastfeeding
* Not taking medications known to cause gingival enlargement

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old, older than 70 years old
* Smokers/tobacco users
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Patients that have severe gingival recession (Miller class III and IV) or < 2 mm.
* Presence of periodontal disease at the recipient site.
* Poor oral hygiene
* Patient pregnant or breastfeeding
* Taking medications known to cause gingival enlargement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unversity of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
Started | 18 | 18 | 18 | 18
Completed | 18 | 18 | 18 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent | Total
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 10 | 6 | 15 | 12 | 43
  >=65 years | 7 | 12 | 3 | 6 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 10 | 10 | 45
  Male | 7 | 4 | 8 | 8 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 17 | 17 | 16 | 15 | 65
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment (0=No Pain to 10=Worst)
Description: To assess the pain outcomes using the visual analog scale from 0=No pain to 10=worst, excrutiating pain. Assessed daily from days 1 to 14, Day 14 reported.
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale | 4.2 (2.4) | 1.9 (2.1) | 2.2 (2.5) | 1 (1.4)

2. Primary Outcome: Bleeding Assessment
Description: To assessed the bleeding outcomes using the visual analog scale (VAS) from 0=No bruising/bleeding to 10=severe bruising/bleeding. Assessed daily from days 1 to 14, Day 14 reported.
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale | 1 (1.9) | 0.6 (1.4) | 0.9 (1.9) | 0.7 (1.6)

3. Secondary Outcome: Activity Tolerance
Description: To assess the effects on daily activities using the visual analog scale from 0=No Limitation to 10= Bedrest required. Assessed daily from days 1 to 14, Day 14 reported.
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale | 2.4 (2.4) | 1.5 (2.1) | 1.8 (2.4) | 1.3 (1.8)

4. Secondary Outcome: Amount of Swelling
Description: To assessed the swelling outcomes using the visual scale (VAS) from 0=No swelling to 10=severe swelling. Assessed daily from days 1 to 14, Day 14 reported.
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale | 2.2 (2.4) | 1.3 (1.9) | 1.4 (2) | 1.3 (2)

5. Secondary Outcome: The Need for Painkiller
Description: To assess the needs for the painkiller using the visual analog scale (VAS). (0 = No painkiller needed to 10 = Needed painkiller). Assessed daily from days 1 to 14, Day 14 reported.
Time Frame: day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
Number analyzed (Participants) | 18 | 18 | 18 | 18
score on a scale | 2.1 (2.5) | 2 (2.6) | 2.2 (2.8) | 1.5 (1.8)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Collagen Plug With Sutures | Platelet Rich Fibrin (PRF) | Collagen Plug With Cyanoacrylate (CPC) | Palatal Stent
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03895476/Prot_SAP_000.pdf